CLINICAL TRIAL: NCT04975100
Title: Evaluation of Efficacy and Safety of add-on Sarcosine in Patients With Major Depressive Disorder: A Randomized Controlled Trial
Brief Title: Evaluation of Efficacy and Safety of add-on Sarcosine in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/AIIMSBBSR/PGThesis/21/07
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sarcosine; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The recruited patients will be randomized by block randomization into two treatment groups using computer-generated random codes with an allocation of 1:1. The random allocation code of the participants will be generated by the investigator who will not be involved in patient recruitment. For allocation concealment, sequentially numbered, identical-looking drug dispensing containers will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Patients in the test group will get Sarcosine 500 mg capsules once daily as an add-on to ongoing SSRI treatment.
  Interventions: Drug: Sarcosine and SSRI
- Control (Active Comparator): Patients in the control group will get identical-looking capsules containing placebo in addition to SSRI at an once daily dose
  Interventions: Drug: Placebo and SSRI

INTERVENTIONS:
Drug: Sarcosine and SSRI — Patients in the test group will get Sarcosine 500 mg capsules once daily as an add-on to ongoing SSRI treatment
  Arms: Test
Drug: Placebo and SSRI — Patients in the control group will get identical-looking capsules containing placebo in addition to SSRI at an once daily dose
  Arms: Control

SUMMARY:
One-third of the patients with major depressive disorder do not respond to conventional antidepressants that act through the mono-aminergic system. The available treatment modalities, including SSRIs, are slow to act and have a lag time before showing improvement in symptoms of patients. To overcome these treatment hurdles, add-on therapy to standard antidepressant drugs may lead to better therapeutic outcomes. Sarcosine, which is a nutraceutical, modulates glutamate neurotransmission has an ameliorative effect on the disease symptoms of depression and negative symptoms of schizophrenia. The only clinical study done on depressive patients by Huang et al. cannot be generalized due to certain inherent limitations. To date, there is no randomized controlled trial with add-on sarcosine to current antidepressant therapy to the best of our knowledge. So, we considered sarcosine can be the candidate drug for add-on therapy due to its multiple mechanisms on the glutaminergic system. Adding sarcosine to ongoing antidepressant therapy may either increase their response rate or decrease adverse drug reactions by decreasing the dose requirement or may show a quicker therapeutic effect. Hence, the present randomized controlled trial has been planned to evaluate the efficacy and safety of sarcosine as add-on therapy in major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder or unipolar depression is a commonly encountered psychiatric disorder, with reported lifetime and one-year prevalence rates of 16.6% and 6.6%, respectively, and is associated with an increased risk of suicide. It is estimated that more than 264 million of the global population have suffered from depression. Major depressive disorder causes significant disabilities, thus adversely affects the quality of life of patients and their caregivers. Despite the clinical significance of depression, its underlying pathophysiology is still not understood comprehensibly, and different potential targets have been explored. One of the most well-researched theories of previous decades has been the monoamine hypothesis; however, it appears that simple monoamine depletion is insufficient to account for the development of the disorder. Drugs acting through enhancing the monoaminergic pathway, i.e., increasing the synaptic concentration of serotonin, noradrenaline, or dopamine, are the most commonly prescribed antidepressant medication in the last five decades. Among them, second-generation antidepressant drugs like selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs) are the most effective and most widely used nowadays.

N-Methyl D-Aspartate receptor (NMDAR) modulation is one of the leading novel mechanisms in the pathophysiology of depression that has been postulated for the treatment of depression. The NMDA hypothesis originated from an unexpected observation that D-cycloserine, a partial agonist of the NMDAR, has antidepressant activity. Also, NMDA-enhancing treatment results in a significant reduction in depressive symptoms in patients with schizophrenia. It has also been observed that major depression is associated with decreased expression and release of brain-derived neurotrophic factors (BDNF).

Sarcosine (N-Methyl Glycine), an endogenous amino acid with NMDA receptor function enhancing property, is usually used as a dietary supplement or nutraceutical. Sarcosine increases the availability of glycine for the glycine binding site of the NMDA receptor by inhibiting its reuptake from the synaptic cleft. It also possesses glycine binding site co-agonistic activity. In various animal studies, it has been found that long-term sarcosine treatment significantly ameliorated the induced depression, confirming the potential role of sarcosine as an antidepressant agent. Huang et al. and Chen et al. have demonstrated antidepressant effects of sarcosine in animal behavior models of depression. The only clinical trial of sarcosine done on depressive patients by Huang et al. has shown better and quicker response with superior tolerability as compared to citalopram.

Therapeutic latency, lack of efficacy in a significant proportion of patients, and adverse drug reactions are the primary concerns in current antidepressant therapies. To overcome these treatment challenges, add-on therapy to standard antidepressant drugs may lead to better therapeutic outcomes. Our literature search found that to date, there is no randomized controlled trial on sarcosine as an add-on therapy to first-line antidepressants like SSRIs. The result of the previous study by Huang et al. cannot be generalized because of the inherent limitations in study design. So, the present randomized controlled trial has been planned to evaluate the efficacy and safety of add-on sarcosine to SSRIs in major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years, of either gender with the clinical diagnosis of major depressive disorder (DSM 5).
* Patients with MADRS score ≥ 7 and ≤ 34 (Mild to moderate severity).
* Patients who are on a stable dose of Sertraline 50 mg or any other SSRI (selective serotonin reuptake inhibitor) therapy in equivalent dose.
* Patients who have given informed written consent.

Exclusion Criteria:

* Major depressive patient treated with Electro Convulsive Therapy recently.
* History of epilepsy, head trauma, or other major neurological or medical disorders.
* Patients with a history of bipolar depression.
* Patients with schizophrenia or other psychotic disorder.
* Patients with suicidal risk.
* Patients with cognitive impairment.
* Initiating or stopping formal psychotherapy within six weeks before enrolment.
* Patients with comorbidities like any malignancies, hepatic, renal, cardiovascular, neurological or endocrinal, respiratory dysfunction.
* Substance abuse history of psychoactive agents.
* Pregnant and lactating mothers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in severity of depressive symptoms from baseline. | 8 weeks
  The change in symptoms of depression will be evaluated using Montgomery Asberg Depression Rating Scale score. Each item of the questionnaire yields a score of 0 to 6. The overall score ranges from 0 to 60. A higher score indicates more severe depression.

SECONDARY OUTCOMES:
Response rate | 8 weeks
  Response rate is defined by percentage of patients showing 50% decrease in MADRS scores from baseline.
Remission rate | 8 weeks
  Remission rate is defined by percentage of patients achieving MADRS scores <7 at 8-week follow-up.
Severity of symptoms | Baseline
  Severity of symptoms at baseline will be assessed by Clinical Global Impression severity scale. The Clinical Global Impression Severity scale is a 7-point scale that requires the clinician to rate the severity of the patient's illness. A higher score reflects more severe illness.
Change in severity of symptoms | 8 weeks
  Change in severity of symptoms will be assessed by Clinical Global Impression Improvement scale. The Clinical Global Impression Improvement scale is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. A lower value reflects better improvement of symptoms.
Change in serum Brain Derived Neurotrophic Factor (BDNF) from baseline | 8 weeks
  Serum BDNF levels will be measured using a commercially available human enzyme-linked immunosorbent assay (ELISA) kit.
Change in serum Glycine from baseline | 8 weeks
  Serum Glycine levels will be measured using a commercially available human enzyme-linked immunosorbent assay (ELISA) kit.
Incidence of adverse drug reactions | 8 weeks
  During the follow-up visit, occurrence of adverse events will be assessed by the nondirective questioning to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, MD, Study Chair — AIIMS, Bhubaneswar
Locations (1):
- AIIMS, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided later.

REFERENCES:
- [Result] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Result] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Result] Hawton K, van Heeringen K. Suicide. Lancet. 2009 Apr 18;373(9672):1372-81. doi: 10.1016/S0140-6736(09)60372-X. PMID 19376453
- [Result] Hasler G. Pathophysiology of depression: do we have any solid evidence of interest to clinicians? World Psychiatry. 2010 Oct;9(3):155-61. doi: 10.1002/j.2051-5545.2010.tb00298.x. PMID 20975857
- [Result] Ruhe HG, Mason NS, Schene AH. Mood is indirectly related to serotonin, norepinephrine and dopamine levels in humans: a meta-analysis of monoamine depletion studies. Mol Psychiatry. 2007 Apr;12(4):331-59. doi: 10.1038/sj.mp.4001949. Epub 2007 Jan 16. PMID 17389902
- [Result] Perez-Caballero L, Torres-Sanchez S, Romero-Lopez-Alberca C, Gonzalez-Saiz F, Mico JA, Berrocoso E. Monoaminergic system and depression. Cell Tissue Res. 2019 Jul;377(1):107-113. doi: 10.1007/s00441-018-2978-8. Epub 2019 Jan 10. PMID 30627806
- [Result] Pochwat B, Nowak G, Szewczyk B. An update on NMDA antagonists in depression. Expert Rev Neurother. 2019 Nov;19(11):1055-1067. doi: 10.1080/14737175.2019.1643237. Epub 2019 Jul 22. PMID 31328587
- [Result] Phillips C. Brain-Derived Neurotrophic Factor, Depression, and Physical Activity: Making the Neuroplastic Connection. Neural Plast. 2017;2017:7260130. doi: 10.1155/2017/7260130. Epub 2017 Aug 8. PMID 28928987
- [Result] Lee MY, Lin YR, Tu YS, Tseng YJ, Chan MH, Chen HH. Effects of sarcosine and N, N-dimethylglycine on NMDA receptor-mediated excitatory field potentials. J Biomed Sci. 2017 Feb 28;24(1):18. doi: 10.1186/s12929-016-0314-8. PMID 28245819
- [Result] Peyrovian B, Rosenblat JD, Pan Z, Iacobucci M, Brietzke E, McIntyre RS. The glycine site of NMDA receptors: A target for cognitive enhancement in psychiatric disorders. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Jun 8;92:387-404. doi: 10.1016/j.pnpbp.2019.02.001. Epub 2019 Feb 6. PMID 30738126
- [Result] Chen KT, Wu CH, Tsai MH, Wu YC, Jou MJ, Huang CC, Wei IH. Antidepressant-like effects of long-term sarcosine treatment in rats with or without chronic unpredictable stress. Behav Brain Res. 2017 Jan 1;316:1-10. doi: 10.1016/j.bbr.2016.06.004. Epub 2016 Aug 21. PMID 27555541
- [Result] Huang CC, Wei IH, Huang CL, Chen KT, Tsai MH, Tsai P, Tun R, Huang KH, Chang YC, Lane HY, Tsai GE. Inhibition of glycine transporter-I as a novel mechanism for the treatment of depression. Biol Psychiatry. 2013 Nov 15;74(10):734-41. doi: 10.1016/j.biopsych.2013.02.020. Epub 2013 Apr 3. PMID 23562005
- [Result] Commons KG, Linnros SE. Delayed Antidepressant Efficacy and the Desensitization Hypothesis. ACS Chem Neurosci. 2019 Jul 17;10(7):3048-3052. doi: 10.1021/acschemneuro.8b00698. Epub 2019 Mar 11. PMID 30807103
- [Result] Chen KT, Tsai MH, Wu CH, Jou MJ, Wei IH, Huang CC. AMPA Receptor-mTOR Activation is Required for the Antidepressant-Like Effects of Sarcosine during the Forced Swim Test in Rats: Insertion of AMPA Receptor may Play a Role. Front Behav Neurosci. 2015 Jun 18;9:162. doi: 10.3389/fnbeh.2015.00162. eCollection 2015. PMID 26150775
- [Derived] Padhan M, Mohapatra D, Mishra BR, Maiti R, Jena M. Efficacy and safety of add-on sarcosine in patients with major depressive disorder: A randomized controlled trial. J Psychiatr Res. 2024 Oct;178:298-304. doi: 10.1016/j.jpsychires.2024.08.026. Epub 2024 Aug 22. PMID 39180989